CLINICAL TRIAL: NCT07332078
Title: Evaluating the Impact of a Low-Cost Food Storage Cabinet ("Meatsafe") on Complementary Food Contamination and Diarrheal Disease in Low-Income Urban Households: A Randomized Controlled Trial in Dhaka, Bangladesh
Brief Title: Meatsafe Food Storage and Diarrhea Prevention Trial in Urban Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 092000310-UCB-0310
Record Dates: First submitted 2025-11-18; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Diarrhea
Keywords: Food Safety; Complementary Foods; Food Hygiene; Safe Food Storage; Meatsafe; Bangladesh; Urban Slum; Low- and Middle-Income Countries (LMICs); WASH (Water, Sanitation, and Hygiene); Enteric Pathogens; Randomized Controlled Trial (RCT); Low-Cost Intervention; Complementary Feeding; Public Health Intervention; Foodborne Pathogens; Enteric Infection; Diarrheal Disease; Fecal-Oral Transmission; Microbial Contamination; Foodborne Illness; Childhood Diarrhea Prevention; Child Health; Escherichia coli (E. coli); Nutrition; Hygiene
MeSH Terms: conditions — Diarrhea; Foodborne Diseases; Escherichia coli Infections

STUDY DESIGN:
Intervention Model Description: Two-arm RCT in which households were randomly allocated to receive either no intervention (control) or a meatsafe with food storage education (intervention).
Masking Description: Not applicable. The intervention is visible (physical food storage cabinet called meatsafe), and masking is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Meatsafe Arm (Experimental): Households received a low-cost, mesh-covered food storage cabinet ("meatsafe") and one-time, in-person education on safe food storage and hygiene. Caregivers also received an illustrated handout to display in the home.
  Interventions: Device: Meatsafe Food Storage Cabinet
- Control Arm (No Intervention): Households did not receive a meatsafe or safe storage education and continued their usual food preparation and storage practices.

INTERVENTIONS:
Device: Meatsafe Food Storage Cabinet — A wire-mesh cabinet for storing cooked food. Designed to prevent contamination from flies, dust, animals, and handling. Distributed with an educational handout and verbal instruction on safe food storage.
  Arms: Intervention Meatsafe Arm

SUMMARY:
The goal of this clinical trial was to evaluate whether a simple household food storage cabinet called a "meatsafe" could reduce bacterial contamination of complementary foods and decrease diarrhea among children aged 6 to 24 months living in low-income settlements of Dhaka, Bangladesh.The study compared households that received a meatsafe and one-time food storage education with households that continued their usual practices. Participating caregivers completed surveys; provided stored food samples for microbiological testing; answered questions about recent child illness; and took part in spot checks of household hygiene and meatsafe use. The trial generated evidence on whether a low-cost and practical tool could help keep children's food safer and reduce diarrheal disease in settings without reliable refrigeration.

DETAILED DESCRIPTION:
Diarrhea remained a major cause of illness and death among children under five years old in low- and middle-income countries (LMICs). In Bangladesh, complementary foods for young children were frequently contaminated with Escherichia coli (E. coli). Storing food uncovered exposed it to contamination from flies, dust, animals, and hands. Existing water, sanitation, and hygiene (WASH) programs did not directly address food hygiene within the home. This randomized controlled trial (RCT) tested whether a low-cost, mesh-covered food storage cabinet ("meatsafe") could reduce microbial contamination of cooked food in urban settlements in Dhaka. Meatsafes were commercially available in local markets and familiar to many households. A total of 290 households living in the Mirpur and Korail settlements were enrolled. Each household had at least one child aged 6 to 24 months. The protocol originally anticipated enrolling 252 households, but 290 were enrolled to maintain balanced allocation and mitigate attrition. Households were randomly assigned to the intervention or control group. Study staff completed follow-up visits every two weeks through Week 10 (five post-intervention follow-ups). Households in the control group did not receive a meatsafe or food hygiene education and continued their usual food storage practices. Households in the intervention group received a free meatsafe and one-time, in-person education on safe food storage and hygiene, along with an illustrated handout to display in the home. Participating households completed surveys on demographics, hygiene behaviors, child feeding, and health; provided stored food samples that were tested for E. coli using culture plating with colony-forming units per gram (CFU/g) enumeration; reported any child diarrhea in the previous seven days; and participated in spot checks of household hygiene and meatsafe use. The primary outcome was the prevalence of complementary food samples with >= 100 CFU/g of E. coli. Secondary outcomes included caregiver-reported diarrhea, dietary diversity, snack and street-food consumption, and measures of meatsafe use and functionality. This study produced evidence on whether providing meatsafes could improve food safety and reduce diarrheal disease among young children in dense urban communities.

ELIGIBILITY:
Inclusion Criteria:

* Household had at least one child aged 6 to 24 months.
* Adult caregiver aged 18 years or older, responsible for child feeding, provided informed consent.
* Household had lived in the study area for at least 6 months and expected to remain for at least 6 additional months.
* Caregiver demonstrated willingness to comply with the assigned intervention or control.

Exclusion Criteria:

* Household owned a functional meatsafe or refrigerator.
* Household planned relocation outside the study area within 6 months.
* Caregiver did not provide informed consent.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 290 (Actual)
Dates: Start 2024-08-11 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of high-level E. coli contamination (>=100 colony-forming units per gram of food, cfu/g) in complementary food samples | Baseline; Weeks 2, 4, 6, 8, and 10
  Food samples were collected from stored complementary foods and tested using standard culture plating. Colony counts were recorded as colony-forming units per gram (CFU/g). Samples with >=100 CFU/g were classified as unsafe per international microbiological standards.
  Safety Issue: No

SECONDARY OUTCOMES:
7-day caregiver-reported diarrhea in children less than 23 months old | Baseline; Weeks 2, 4, 6, 8, and 10
  Diarrhea was defined per World Health Organization (WHO) criteria as >=3 loose stools within a 24-hour period in the past 7 days.
Duration of food storage | Weeks 2, 4, 6, 8, and 10
  Data collectors will record the duration that prepared complementary foods are stored using the following defined categories: <=4 hours, >4 to 8 hours and >8 hours.
Temperature of food storage location | Weeks 2, 4, 6, 8, and 10
  Ambient temperature of the food storage area was measured in degrees Celsius using a digital thermometer.
Humidity of food storage location | Weeks 2, 4, 6, 8, and 10
  Relative humidity of the food storage environment was recorded as a percentage (%) using a digital hygrometer.
Recall of food hygiene and meatsafe behavior-change messages | Week 10
  Caregivers were asked to recall and describe key hygiene and storage messages from the educational handout.
Meatsafe functionality | Weeks 2, 4, 6, 8, and 10.
  Spot checks observation of functionality of the food storage cabinet assessed using a 3-category rating: does not close / difficult to close / closes easily. These categories do not represent a numerical or ordinal scale.
Meatsafe Cleanliness | Weeks 2, 4, 6, 8, and 10
  Spot checks observation of cleanliness assessed using a 3-category rating: considerable dirt / some dirt / very clean. These categories do not represent a numerical or ordinal scale.
Meatsafe screen condition | Weeks 2, 4, 6, 8, and 10
  Spot checks observation of screen condition assessed using a 3-category rating: multiple holes / one hole / no holes. These categories do not represent a numerical or ordinal scale.

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including household survey responses and microbiological food sample results, may be shared upon reasonable request. Only de-identified data will be shared, with all personal identifiers removed, and use will be consistent with participant consent and approvals by the relevant institutional review boards: UC Berkeley Committee for Protection of Human Subjects (CPHS) and icddr,b Ethical Review Committee (ERC).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months after publication of primary findings and continuing for 3 years.
Access Criteria: Researchers with a methodologically sound proposal may request access to de-identified IPD and supporting documents. Requests must be reviewed and approved by the principal investigators and the relevant institutional review boards (UC Berkeley CPHS and icddr,b ERC). Data will be shared under a data use agreement and transferred through secure systems.